CLINICAL TRIAL: NCT04876430
Title: Open-label Randomized Clinical Trial Comparing Best Available Therapy With or Without Meropenem for Bloodstream Infections by Enterobacterales With Minimal Inhibitory Concentrations for Meropenem Above 32mg/L
Brief Title: Best Available Therapy With or Without Meropenem for Bloodstream Infections by Enterobacterales With High Level of Resistance to Carbapenems
Acronym: ABOVE
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Very low frequency of recruitment
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Collaborators: Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government)
Responsible Party: Principal Investigator, Alexandre Prehn Zavascki, Principal Investigator, Hospital de Clinicas de Porto Alegre
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2019-0401
Record Dates: First submitted 2021-05-03; First posted 2021-05-06 (Actual); Last update posted 2022-08-03 (Actual); Status verified 2022-08

CONDITIONS: Carbapenem-Resistant Enterobacteriaceae Infection; Bloodstream Infection
Keywords: carbapenem; carbapenemase; polymyxins; treatment; carbapenem resistance
MeSH Terms: conditions — Sepsis | interventions — Meropenem

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Meropenem plus Best Available Therapy plus (Experimental): Meropenem 2g every 8 hours combined with the best available therapy (BAT). BAT will be defined according to the susceptibility profile and decision of the assistant team before randomization and should include at least one of the antimicrobials that, usually, have in vitro activity against carbapenem-resistant Enterobacterales isolates.
  1. Polymyxin B or colistimethate;
  2. Amikacin or gentamicin;
  3. Tigecycline;
  4. Another antimicrobial with in vitro susceptibility.
  Doses will be defined by the assistant team.
  Interventions: Drug: Meropenem
- Best Available Therapy (No Intervention): The best available therapy will be defined according to the susceptibility profile and decision of the assistant team before randomization and should include at least one of the antimicrobials that, usually, have in vitro activity against carbapenem-resistant Enterobacterales isolates.
  1. Polymyxin B or colistimethate;
  2. Amikacin or gentamicin;
  3. Tigecycline;
  4. Another antimicrobial with in vitro susceptibility.
  Doses will be defined by the assistant team.

INTERVENTIONS:
Drug: Meropenem — Meropenem 2g every 8h for patients with glomerular filtration rate (GFR) equal or higher that 50 mL/min. Dose adjustment is recommended for patients with GFR < 50mL/min.
  Arms: Meropenem plus Best Available Therapy plus

SUMMARY:
Enterobacterales resistant to carbapenem are cause of severe concern in hospital-acquired infections since therapeutic options are limited. Recently approved drugs, such as bela-lactam/beta-lactamase inhibitor, have been the drug of choice. However, its use is limited in low- and middle-income countries. Thus, therapy of these infections mostly relies on polymyxins and other old drugs.

The role of adjuvant carbapenem therapy in combination with polymyxins, aminoglycosides and other drugs is under investigation. From a pharmacokinetic/pharmacodynamic (PK/PD), there is an elevated probability that high-dose, extended infusion administered meropenem reach the PK/PD target of 40% above the minimal inhibitory concentration (MIC) of the pathogen when the MIC is 32mg/L or lower (non-susceptible isolates have MICs of 4mg/L or higher). However, the MIC is not routinely determined in clinical laboratories. In addition, high-level (above 32mg/L) resistance to carbapenems have been reported in many studies.

This open-label, randomized clinical trial aim to assess if the addition of meropenem to the best available therapy can increase the number of days alive and free of hospitalization in patients with bloodstream infections by Enterobacterales with MIC of meropenem above 32mg/L.

ELIGIBILITY:
Inclusion Criteria:

* Primary or secondary bloodstream infections by any specie of the Enterobacterales family with minimum inhibitory concentration (MIC) for meropenem >32mg/L;
* Agreement of the assistant team with the inclusion of the patient in the study;
* Agreement by the patient or legal guardian to sign the informed consent form.

Exclusion Criteria:

* Known pregnancy;
* Patients belonging to the population deprived of their liberty;
* Known allergy to meropenem;
* Use of ceftazidime-avibactam (or any other new antimicrobial agent that become available in Brazil during the study period) for the treatment of the current infection;
* Infection by an Enterobacterales isolates without in vitro susceptibility to at least one antimicrobial drug;
* Bloodstream co-infection by another gram negative bacilli;
* Concomitant infection at any site by a pathogen which meropenem is indicated;
* Neutropenia (<1000 neutrophils cells/mm3)
* Death expected within 48 hours of eligibility assessment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2021-05-04 (Actual); Primary Completion 2022-03-07 (Actual); Study Completion 2022-03-07 (Actual)

PRIMARY OUTCOMES:
Days alive and free of hospitalization | 60 days
  Number of days in which patients are alive and out of the hospital

SECONDARY OUTCOMES:
Overall mortality | 14, 28 and 60 days after randomization
  Death for any cause
Antimicrobial-free days | 60 days after randomization
  Number of days in which patients are alive and without use of antimicrobial drugs
Relapse of infection | 60 days after randomization
  Presence of infection with isolation of the same bacteria between 14 and 60 days after randomization.
Clostridioides difficile infection | 60 days after randomization
  Incidence of Clostridioides difficile infection
Acute Kidney Injury | 14 days after randomization
  Incidence of Acute Kidney Injury, according to Kidney Disease: Improving Global Outcomes (KDIGO) criteria
Meropenem-related adverse effects | 14 days after randomization
  Incidence of adverse effects related to meropenem, such as neurological toxicity and hypersensitivity reactions

CONTACTS AND LOCATIONS:
Locations (2):
- Brazil (2):
  - Hospital de Clínicas de Porto Alegre, Porto Alegre, Rio Grande do Sul
  - Hospital São Lucas da Pontifícia Universidade Católica do Rio Grande do Sul, Porto Alegre, Rio Grande do Sul